CLINICAL TRIAL: NCT03472482
Title: Optical Coherence Tomography in Cerebral Amyloidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S59048
Record Dates: First submitted 2018-01-19; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer Disease; Dementia Alzheimers; Dementia; Lewy Body Disease; Dementia, Lewy Body; Mild Cognitive Impairment
Keywords: Alzheimer's disease; Dementia; Lewy body disease; Retina; Retinal imaging; Optical Coherence Tomography; Hyperspectral imaging; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Lewy Body Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Ab+ cognitively intact volunteers: amyloid-positive cognitively intact controls (55-80 years)
  interventions: non-invasive retinal imaging with Optical Coherence Tomography (OCT), OCT-angiography (OCT-A), Autofluorescence, Fundus Photography, Hyperspectral Imaging
  Interventions: Diagnostic Test: non-invasive retinal imaging
- Ab- cognitively intact volunteers: amyloid-negative cognitively intact controls (55-80 years)
  interventions: non-invasive retinal imaging with Optical Coherence Tomography (OCT), OCT-angiography (OCT-A), Autofluorescence, Fundus Photography, Hyperspectral Imaging
  Interventions: Diagnostic Test: non-invasive retinal imaging
- amyloid-positive MCI patients: amyloid-positive patients with Mild Cognitive Impairment
  interventions: non-invasive retinal imaging with Optical Coherence Tomography (OCT), OCT-angiography (OCT-A), Autofluorescence, Fundus Photography, Hyperspectral Imaging
  Interventions: Diagnostic Test: non-invasive retinal imaging
- amyloid-negative MCI patients: amyloid-negative patients with Mild Cognitive Impairment
  interventions: non-invasive retinal imaging with Optical Coherence Tomography (OCT), OCT-angiography (OCT-A), Autofluorescence, Fundus Photography, Hyperspectral Imaging
  Interventions: Diagnostic Test: non-invasive retinal imaging
- AD patients: patients in the dementia stage of Alzheimer's Disease
  interventions: non-invasive retinal imaging with Optical Coherence Tomography (OCT), OCT-angiography (OCT-A), Autofluorescence, Fundus Photography, Hyperspectral Imaging
  Interventions: Diagnostic Test: non-invasive retinal imaging
- LBD patients: patients with Lewy Body Dementia
  interventions: non-invasive retinal imaging with Optical Coherence Tomography (OCT), OCT-angiography (OCT-A), Autofluorescence, Fundus Photography, Hyperspectral Imaging
  Interventions: Diagnostic Test: non-invasive retinal imaging

INTERVENTIONS:
Diagnostic Test: non-invasive retinal imaging

SUMMARY:
In this observational study, the investigators aim to evaluate whether changes in the retinal and choroidal circulation, as assessed by Optical Coherence Tomography (OCT) and the quantification of retinal amyloid deposits using auto-fluorescence and hyperspectral retinal imaging, are correlated with the degree and subtype of dementia and with the presence or absence of a positive amyloid scan.

For this purpose, patients with established Alzheimer's Disease (AD) and Lewy Body Dementia (LBD), as well as amyloid positive and amyloid negative Mild Cognitive Impairment (MCI) and aged matched cognitively intact patients will be included in this cross-sectional study.

DETAILED DESCRIPTION:
Being a direct extension of the central nervous system and the only place in the human body where the vessels of the central circulation can be visualized directly, the eye provides a unique window to investigate the central circulatory system. Several studies have demonstrated that retinal blood vessels show structural and functional alterations in patients with dementia. These measurements are based on fundus pictures and are hence limited to the larger retinal vessels.

Until recently, intravenous injection of a contrast agent was necessary to visualize the retinal microvasculature in detail. While indispensable for the diagnosis of some ocular vascular diseases (arterial/venous occlusion, neovascularization,…) the invasiveness of fluorescein angiography (and the risk of an allergic reaction) limits its use as a screening tool to detect alterations in the microvascular network of the retina and choroid.

Optical coherence tomography (OCT) is a non-invasive diagnostic tool capable of generating cross-sectional coupes of the retina and choroid. Novel algorithms allow to render a 3-dimensional model of the ocular microcirculation based merely on the motion contrast of the circulating blood. Since OCT is fast, easy to perform and completely non-invasive, this technique lends itself for screening purposes.

Auto-fluorescence retinal imaging is an imaging modality that is commonly used in ophthalmological practice to assess retinal pigment epithelium and photoreceptor function by quantifying the relative amount of auto-fluorescent lipofuscin. The images can be acquired using the OCT device but require pupil dilation. Using visible light of 488nm, it is a safe imaging technique with no short or late term side-effects to the patient. A recent study has described abnormal auto-fluorescence patterns in patients with cerebral amyloid deposition.

Hyperspectral fundus photography is comparable to regular fundus photography but uses an image sensor that can acquire images at multiple different wavelengths (unlike the classical red-green-blue colour sensors that are used in conventional cameras). Apart from a different image sensor, the device is identical to a regular fundus camera. Recent studies have emerged that describe a unique hyperspectral signature of aggregated retinal amyloid deposits.

The proposed study aims to investigate whether retinal or choroidal vascular parameters measured using OCT and the quantification of retinal amyloid deposits using auto-fluorescence and hyperspectral retinal imaging, could be useful to identify different subpopulations of cognitive intact, MCI and dementia patients.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively intact healthy controls will be recruited from an ongoing community-recruited longitudinal cohort of cognitively intact older adults (55-85 years, S51125) who all have undergone amyloid Positron Emission Tomography (PET) at the baseline visit in the context of study S51125. Half of the subjects will be amyloid-positive and half will be amyloid-negative. In the context of study S51125 these subjects receive two-yearly neuropsychological assessment.
* MCI patients (Petersen et al., 2004 criteria) will be recruited from an ongoing memory-clinic recruited longitudinal cohort of patients with amnestic mild cognitive impairment who participate in study S55892. All subjects have undergone an amyloid PET at the baseline study in the context of study S55892. Half of the subjects will be amyloid-positive and half will be amyloid negative.
* Clinically probable AD subjects (National Institute of Neurological Disorders and Stroke (NINDS) and the Association Internationale pour la Recherche et l'Enseignement en Neurosciences (AIREN) criteria) will be recruited from the memory clinic University Hospitals Leuven (MMSE 12-28). Subjects will be recruited only if they are capable of providing written informed consent.
* Clinically probable LBD (McKeith et al. criteria, 2005) will be recruited from the memory clinic University Hospitals Leuven (MMSE 12-28). Subjects will be recruited only if they are capable of providing written informed consent.
* Capable and willing to participate

Exclusion Criteria:

* Personal medical history of retinal neovascularization
* Unable or unwilling to give consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cfr. Eligibility Criteria
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2016-03-25 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of OCT measurements in dementia | 2 years
  area under the curve (AUC) on receiver operating characteristic curves

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Vandewalle, MD PhD, Principal Investigator — UZ Leuven/KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2016-04-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT03472482/Prot_000.pdf